CLINICAL TRIAL: NCT06391567
Title: Determination of Balance Characteristics in People With Frozen Shoulders
Brief Title: Balance in People With Frozen Shoulder
Status: Completed | Type: Observational
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Atahan TURHAN, Dr. Lecturer, Kirsehir Ahi Evran Universitesi
Other Study IDs: KAEU-T.ATAHAN-002
Record Dates: First submitted 2024-04-18; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Frozen Shoulder
Keywords: Adhesive Capsulitis; Balance; Pain
MeSH Terms: conditions — Bursitis; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group: The control group consisted of healthy subjects who were not diagnosed with Frozen Shoulder and did not have a chronic disease that would affect balance between the ages of 40-65.
  Interventions: Other: There was no intervention in this study.
- Patient Group: Patients who were diagnosed with Frozen Shoulder by physical examination, met the inclusion criteria, and agreed to participate in the study were selected for the patient group.
  Interventions: Other: There was no intervention in this study.

INTERVENTIONS:
Other: There was no intervention in this study. — There was no intervention in this study.

SUMMARY:
The aim of this study was to investigate the balance characteristics of patients with Frozen Shoulder.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers aged 40-65 years,
* Diagnosed with unilateral Frozen Shoulder, Frozen Shoulder stage 2-3,
* Pain lasting more than 3 months,
* No mental or cognitive impairment
* At least 25% movement limitation in at least 2 movement planes and
* Able to cooperate.

Exclusion Criteria:

* Who had a neurological, rheumatic, cardiac and active malignant diseases
* Who had a history of surgery, trauma, and fracture
* Who had comorbid conditions that would affect balance

The control group consisted of healthy subjects who were not diagnosed with Frozen Shoulder and did not have a chronic disease that would affect balance between the ages of 40-65.

Ages: 40 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the Physical Medicine and Rehabilitation Outpatient Clinic with complaints of shoulder pain were examined by a physiatrist. Patients who were diagnosed with Frozen Shoulder by physical examination, who met the inclusion criteria, and who agreed to participate in the study were included in the study. The control group consisted of hospital and university staff. The control group was also assessed by the same physiatrist and confirmed by the country's health database as having no chronic disease affecting balance.
Sampling Method: Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2024-04-10 (Actual); Study Completion 2024-04-16 (Actual)

PRIMARY OUTCOMES:
Sociodemographic Form | 8 week
  Sociodemographic information of the patients included in the study, such as age, gender, height, weight, BMI, educational status, dominant side, comorbid status, and clinical information such as affected side, pain intensity, and pain duration were collected in a case report form by face-to-face interview
Balance Function | 8 week
  Balance function was measured with the Timed Up and Go Test (TUG). The TUG is a short, simple, and reliable test used to assess balance. It shows that people who complete the test in less than 20 seconds are independent in transfers, while people who complete the test in 30 seconds or more are more dependent in activities of daily living.
Static and Dynamic Postural Balance | 8 week
  Biodex Balance System was used for objective assessment of static and dynamic postural balance. A high balance score indicates poor balance performance.
Pain Intensity | 8 week
  The pain intensity of the patients was measured using the Visual Analogue Scale. The pain intensity score ranges from 0 to 10. An increase in the score indicates an increase in pain; a decrease in the score indicates a decrease in pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Atahan TURHAN, Kırşehir, Merkez, Turkey (Türkiye)